CLINICAL TRIAL: NCT05724147
Title: The Effect of Mandala Activity on Happiness and Well-Being Levels in Elderly People Living in Nursing Homes: Colorize Life Project
Brief Title: Mandala Activity in Elderly People Living in Nursing Homes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Atlas University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AtlasU3
Record Dates: First submitted 2023-01-27; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Happiness; Well-being; Older; Elderly
Keywords: Mandala; Older; Elderly; Happiness; Well-being

STUDY DESIGN:
Intervention Model Description: in a single group pretest-posttest research design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mandala Activity (Experimental): There will be a total of 5 sessions, including the Mandala activity once a week, meeting (1), working (3) and ending (1).
  Interventions: Behavioral: Mandala Activity

INTERVENTIONS:
Behavioral: Mandala Activity — Three sessions of mandala activity, once a week, will be applied to the participants from the elderly people in the nursing home included in the study. The mandala activity planned to be done with the group will be done in addition to the standard monitoring applied in the institution, so it will be held at an appropriate time according to the flow in the institution. Before leaving the individuals, the most appropriate time for the next mandala session will be determined by taking into account the preferences of the individuals. Individuals to be included in the study will be grouped in groups of 10. Mandala activity application time is planned to last approximately 2 hours. If individuals have any physical symptoms, the time of the mandala activity is rescheduled, and each individual is expected to attend five sessions during the total study period.

SUMMARY:
The Effect of Mandala Activity on Happiness and Well-Being Levels in Elderly People Living in Nursing Homes: Colorize Life Project

DETAILED DESCRIPTION:
In recent years, there has been a global increase in the elderly population. Biopsychosocial regressions and various health problems are seen in the elderly, and their care and follow-up mostly continue with hospitalization in nursing homes. In studies examining the opinions of elderly individuals staying in nursing homes about the institution they stay, it has been stated that individuals see the institution as an area for making friends and socializing with their peers. In Erikson's theory of psychosocial development, it is stated that in the last stage of old age, individuals experience hopelessness against self-integrity. If his evaluation of his life is positive, self-integrity is achieved, if it is negative, he falls into despair, experiences dissatisfaction and becomes unhappy. In this context, various psychosocial interventions are recommended within the scope of protecting and improving mental health in elderly individuals. In the literature, when the studies using mandala were examined, it was found that the effects of the effects on the children and adolescent groups and the effects on the anxiety levels were mostly evaluated. In the international literature, studies evaluating the effect of mandala activity with elderly individuals are limited, and in our country, no study with this sample has been found. This study is unique in terms of evaluating the effect of mandala activity on elderly individuals living in nursing homes in our country. It is a multi-faceted study since the study is carried out with undergraduate students, it is carried out with students from the psychology and nursing departments, as a multidisciplinary, and it will implement the planned activity with elderly individuals who are hospitalized in a nursing home. At the end of the study, it is predicted that the elderly individuals will increase their happiness and well-being. Undergraduate students taking part in the study will also experience doing an experimental study. When considered in the context of Erikson's psychosocial development theory, it is thought that it is important to support the elderly individuals psychosocially in old age, which is the last stage of life. The study is an experimental study designed in a pretest and posttest pattern. The universe of the study; All nursing homes (n=12) in Şişli district will consist of elderly individuals receiving health care services. In the selection of the sample, first of all, the institution where the study will be carried out will be determined by drawing lots among the institutions, and the elderly individuals who meet the inclusion and exclusion criteria will form the sample of the study. Data will be obtained with Personal Information Form (PIF), Happiness Scale and Well-Being Scale. There will be a total of 5 sessions, including the Mandala activity once a week, meeting (1), working (3) and ending (1). In the study, answers will be sought to the question "Is there a difference between the happiness and well-being levels of individuals before and after the Mandala activity?" The analysis of the data will be done using the SPSS 23.0 package program. In the evaluation of the data, descriptive statistics such as frequency distribution, mean and standard deviation will be used to define the sample, two-pair test or Wilcoxon peer test will be used according to the parametric test assumptions for the comparison of the group within itself, and the Chi-square test will be used for the analysis of categorical data. 95% significance level will be used to determine the differences in the analyses. The answers to the open-ended questions will be categorized by the researchers and evaluated as numbers and percentages. As a result of the study, the effect of mandala activity on the happiness and well-being of the elderly will be determined and a contribution will be made to the literature. It is envisaged that the mandala activity applied in this study will guide further studies. In line with the literature information and justification, this study was planned to determine the effect of mandala activity on happiness and well-being levels in elderly individuals living in nursing homes.

ELIGIBILITY:
Inclusion Criteria:

* Being 60 years or older
* Do not speak Turkish
* Continuing hospitalization in the specified institution,
* Ability to hold pencils, draw, paint,
* Not having any neurological and physical disorders (paralysis, rheumatoid arthritis, etc.) in their hands,
* Volunteering to participate in the study

Exclusion Criteria:

* Having a barrier to communication,
* Having a diagnosis of any mental disorder,

Removal Criteria:

* Not attending 2 sessions or more, The development of a medical condition that hinders the intervention process,
* Leaving the institution,
* The participant's right to withdraw from the research at his/her own request or family

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-03-15 (Estimated); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
Happiness | 5 week
  Happiness Scale. It consists of six five-point Likert-type questions: (1) Not at all suitable for me (2) Not suitable for me (3) Somewhat suitable for me (4) Fairly suitable for me (5) Completely suitable for me. The scores that can be obtained from the scale are between 6-30. The higher the score, the higher the happiness level.
Well-Being | 5 week
  Well-Being Scale. Participants are expected to express their opinions on the scale items on a 7-point Likert-type rating, ranging from 1-strongly disagree to 7-strongly agree. A total well-being score can be obtained by summing the scores of all items in the scale. The highest score that can be obtained from the scale is 56, and the lowest score is 8. There is no reverse scored item in the scale. High scores obtained from the scale indicate that the level of well-being of the individual is high.

CONTACTS AND LOCATIONS:
Locations (1):
- Şeyma Demiralay, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
I can share to contribute to the literature
Time Frame: 6 months